CLINICAL TRIAL: NCT03264898
Title: Comparative Effectiveness of Fecal Immunochemical Tests With Optical Colonoscopy (R01 CA215034)
Brief Title: Comparative Effectiveness of FITs With Colonoscopy
Acronym: BestFIT
Status: Completed | Type: Observational
Sponsor: Barcey T. Levy (Other)
Collaborators: University of North Carolina (Other); Texas Tech University Health Sciences Center (Other)
Responsible Party: Sponsor-Investigator, Barcey T. Levy, Professor, University of Iowa
Organization: University of Iowa (Other)
Other Study IDs: IRB ID#201610814
Record Dates: First submitted 2017-08-21; First posted 2017-08-29 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Fecal Immunochemical Test (FIT) Group: Each participant will complete 5 different FITs, on a single stool sample collected in a hat. Each participant will undergo optical colonoscopy and their FIT results compared with their colonoscopy with biopsy results (if applicable). We will calculate the test characteristics of each FIT.
  Interventions: Device: Fecal immunochemical test (FIT)

INTERVENTIONS:
Device: Fecal immunochemical test (FIT) — FIT is a type of fecal occult blood test that uses antibodies to hemoglobin to detect blood in stool.

SUMMARY:
Colorectal cancer is a preventable and/or a treatable cancer, but at least 43% of the United States population is not up-to-date with screening. Although 90% of colorectal cancer screening is done using colonoscopy, most other countries use fecal immunochemical tests, reserving colonoscopy for those with a positive fecal immunochemical test. This project will provide the foundation for a paradigm shift for colorectal cancer screening in the United States by identifying how well 5 different FITs work for detecting screening relevant neoplasia, thus reducing morbidity and mortality for colorectal cancer.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is the third most common cancer and the third leading cause of cancer death in both men and women in the U.S., with nearly 50,000 deaths each year. Since CRC develops over a number of years from precursor lesions called polyps, it is largely detectable and preventable in early stages. As these polyps become larger, they, like most CRCs, tend to bleed, which is the rationale for the use of fecal occult blood tests (FOBTs) to detect both polyps and cancers early, while they are curable. However, early screening and detection is much less common than it could be, with about 43% of eligible individuals unscreened. Fecal immunochemical tests (FITs) are a type of FOBT that can be a sensitive, specific, and low cost alternative to colonoscopy for CRC screening. Modeling studies have shown that for population screening, a strategy of annual FIT testing from age of 50 to 75 years results in an equal number of life-years gained as compared with colonoscopy every 10 years. However, about 90% of screening in the U.S. is done with colonoscopy, the most expensive and invasive screening test. FITs are far less costly and largely replacing the guaiac test in CRC screening programs internationally, where only individuals with positive results are referred for a colonoscopy. Studies done on FITs in other countries often used FITs not available in the U.S. or studied high-risk populations; thus, results are not applicable in the U.S. It is critical to determine the FIT(s) with the best test characteristics in order to implement successful FIT-based screening programs in this country.

It is estimated that 24 million more individuals will need to be screened by 2018 to reach the "80% by 2018" goal set by the National Colorectal Cancer Roundtable. To address this knowledge gap, investigators propose to compare the test characteristics of three Clinical Laboratory Improvement Amendments (CLIA)-waived FITs and two automated FITs, using colonoscopy as the gold standard. The rationale for this proposed study is that, for almost all of the FITs currently marketed in the U.S., there is no evidence of the accuracy claimed. Specific aims are: Aim 1: To assess the diagnostic accuracy for advanced colorectal neoplasms of three of the most commonly used CLIA-waived FITs and two automated FITs, using colonoscopy as the gold standard.

Aim 2: To evaluate the diagnostic accuracy of two quantitative FITs using receiver operating characteristic (ROC) analysis. Aim 3: To assess factors associated with false positive and false negative FIT results for each device.

These findings will provide essential information about FITs with the best test characteristics for future expanded use of FIT, critically important to achieving the long-term goal of reducing morbidity and mortality from CRC. FITs are more acceptable to patients, will allow higher screening rates, and will reduce costs as compared with a screening strategy based on colonoscopy as the primary initial screening method.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for a screening or surveillance colonoscopy

Exclusion Criteria:

* familial polyposis syndromes: ulcerative colitis or Crohn's disease: or active rectal bleeding

Ages: 50 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients being scheduled for screening or surveillance colonoscopies meeting the study criteria at three academic health centers
Sampling Method: Non-Probability Sample
Enrollment: 3761 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
Advanced adenoma or cancer as assessed by colonoscopy with biopsy if needed | About 21 days from collection of FIT to performance of colonoscopy
  Individual FIT brand results of negative, positive, or invalid

CONTACTS AND LOCATIONS:
Overall Officials: Barcey T Levy, PhD, MD, Principal Investigator — University of Iowa
Locations (3):
- United States (3):
  - University of Iowa, Iowa City, Iowa
  - University of North Carolina, Chapel Hill, North Carolina
  - Texas Tech University Health Sciences Center, El Paso, Texas

IPD SHARING:
Plan to Share IPD: Yes
Once the key publications are accepted and finalized, de-identified data and the codebook will be made available to anyone with a legitimate request who follows the Data Sharing agreement.
Time Frame: Once study key publications have been accepted and finalized for publication.
Access Criteria: Researchers have to make a formal proposal for data and codebook.

REFERENCES:
- [Background] Smith RA, Andrews K, Brooks D, DeSantis CE, Fedewa SA, Lortet-Tieulent J, Manassaram-Baptiste D, Brawley OW, Wender RC. Cancer screening in the United States, 2016: A review of current American Cancer Society guidelines and current issues in cancer screening. CA Cancer J Clin. 2016 Mar-Apr;66(2):96-114. doi: 10.3322/caac.21336. Epub 2016 Jan 21. PMID 26797525
- [Background] Kuntz KM, Lansdorp-Vogelaar I, Rutter CM, Knudsen AB, van Ballegooijen M, Savarino JE, Feuer EJ, Zauber AG. A systematic comparison of microsimulation models of colorectal cancer: the role of assumptions about adenoma progression. Med Decis Making. 2011 Jul-Aug;31(4):530-9. doi: 10.1177/0272989X11408730. Epub 2011 Jun 14. PMID 21673186
- [Background] Young GP, Symonds EL, Allison JE, Cole SR, Fraser CG, Halloran SP, Kuipers EJ, Seaman HE. Advances in Fecal Occult Blood Tests: the FIT revolution. Dig Dis Sci. 2015 Mar;60(3):609-22. doi: 10.1007/s10620-014-3445-3. Epub 2014 Dec 10. PMID 25492500
- [Background] Fedewa SA, Sauer AG, Siegel RL, Jemal A. Prevalence of major risk factors and use of screening tests for cancer in the United States. Cancer Epidemiol Biomarkers Prev. 2015 Apr;24(4):637-52. doi: 10.1158/1055-9965.EPI-15-0134. PMID 25834147
- [Background] Robertson DJ, Imperiale TF. Stool Testing for Colorectal Cancer Screening. Gastroenterology. 2015 Oct;149(5):1286-93. doi: 10.1053/j.gastro.2015.05.045. Epub 2015 May 30. PMID 26033632
- [Background] Allison JE. The best screening test for colorectal cancer is the one that gets done well. Gastrointest Endosc. 2010 Feb;71(2):342-5. doi: 10.1016/j.gie.2009.10.032. No abstract available. PMID 20152313
- [Background] Hawley ST, Volk RJ, Krishnamurthy P, Jibaja-Weiss M, Vernon SW, Kneuper S. Preferences for colorectal cancer screening among racially/ethnically diverse primary care patients. Med Care. 2008 Sep;46(9 Suppl 1):S10-6. doi: 10.1097/MLR.0b013e31817d932e. PMID 18725820
- [Background] Wolf RL, Basch CE, Brouse CH, Shmukler C, Shea S. Patient preferences and adherence to colorectal cancer screening in an urban population. Am J Public Health. 2006 May;96(5):809-11. doi: 10.2105/AJPH.2004.049684. Epub 2006 Mar 29. PMID 16571715
- [Background] Xu Y, Levy BT, Daly JM, Bergus GR, Dunkelberg JC. Comparison of patient preferences for fecal immunochemical test or colonoscopy using the analytic hierarchy process. BMC Health Serv Res. 2015 Apr 23;15:175. doi: 10.1186/s12913-015-0841-0. PMID 25902770
- [Background] Zauber AG, Lansdorp-Vogelaar I, Knudsen AB, Wilschut J, van Ballegooijen M, Kuntz KM. Evaluating test strategies for colorectal cancer screening: a decision analysis for the U.S. Preventive Services Task Force. Ann Intern Med. 2008 Nov 4;149(9):659-69. doi: 10.7326/0003-4819-149-9-200811040-00244. Epub 2008 Oct 6. PMID 18838717
- [Background] Zavoral M, Suchanek S, Majek O, Fric P, Minarikova P, Minarik M, Seifert B, Dusek L. Colorectal cancer screening: 20 years of development and recent progress. World J Gastroenterol. 2014 Apr 14;20(14):3825-34. doi: 10.3748/wjg.v20.i14.3825. PMID 24744575
- [Background] Centers for Disease Control and Prevention (CDC). Vital signs: colorectal cancer screening test use--United States, 2012. MMWR Morb Mortal Wkly Rep. 2013 Nov 8;62(44):881-8. PMID 24196665
- [Background] Zavoral M, Suchanek S, Zavada F, Dusek L, Muzik J, Seifert B, Fric P. Colorectal cancer screening in Europe. World J Gastroenterol. 2009 Dec 21;15(47):5907-15. doi: 10.3748/wjg.15.5907. PMID 20014454
- [Background] de Wijkerslooth TR, Stoop EM, Bossuyt PM, Meijer GA, van Ballegooijen M, van Roon AH, Stegeman I, Kraaijenhagen RA, Fockens P, van Leerdam ME, Dekker E, Kuipers EJ. Immunochemical fecal occult blood testing is equally sensitive for proximal and distal advanced neoplasia. Am J Gastroenterol. 2012 Oct;107(10):1570-8. doi: 10.1038/ajg.2012.249. Epub 2012 Jul 31. PMID 22850431
- [Background] Levi Z, Rozen P, Hazazi R, Vilkin A, Waked A, Maoz E, Birkenfeld S, Leshno M, Niv Y. A quantitative immunochemical fecal occult blood test for colorectal neoplasia. Ann Intern Med. 2007 Feb 20;146(4):244-55. doi: 10.7326/0003-4819-146-4-200702200-00003. PMID 17310048
- [Background] Seeff LC, Richards TB, Shapiro JA, Nadel MR, Manninen DL, Given LS, Dong FB, Winges LD, McKenna MT. How many endoscopies are performed for colorectal cancer screening? Results from CDC's survey of endoscopic capacity. Gastroenterology. 2004 Dec;127(6):1670-7. doi: 10.1053/j.gastro.2004.09.051. PMID 15578503
- [Background] Sharara AI, El Reda ZD, Harb AH, Abou Fadel CG, Sarkis FS, Chalhoub JM, Abou Mrad R. The burden of bowel preparations in patients undergoing elective colonoscopy. United European Gastroenterol J. 2016 Apr;4(2):314-8. doi: 10.1177/2050640615594550. Epub 2015 Jul 3. PMID 27087962
- [Background] Imperiale TF, Ransohoff DF, Itzkowitz SH, Levin TR, Lavin P, Lidgard GP, Ahlquist DA, Berger BM. Multitarget stool DNA testing for colorectal-cancer screening. N Engl J Med. 2014 Apr 3;370(14):1287-97. doi: 10.1056/NEJMoa1311194. Epub 2014 Mar 19. PMID 24645800
- [Background] Levy BT, Bay C, Xu Y, Daly JM, Bergus G, Dunkelberg J, Moss C. Test characteristics of faecal immunochemical tests (FIT) compared with optical colonoscopy. J Med Screen. 2014 Sep;21(3):133-43. doi: 10.1177/0969141314541109. Epub 2014 Jun 23. PMID 24958730
- [Background] Levi Z, Rozen P, Hazazi R, Vilkin A, Waked A, Maoz E, Birkenfeld S, Lieberman N, Klang S, Niv Y. Sensitivity, but not specificity, of a quantitative immunochemical fecal occult blood test for neoplasia is slightly increased by the use of low-dose aspirin, NSAIDs, and anticoagulants. Am J Gastroenterol. 2009 Apr;104(4):933-8. doi: 10.1038/ajg.2009.14. Epub 2009 Mar 17. PMID 19293792
- [Background] Crouse AL, De Koning L, Sadrzadeh SM, Naugler C. Sensitivity and Specificity of Community Fecal Immunotesting Screening for Colorectal Carcinoma in a High-Risk Canadian Population. Arch Pathol Lab Med. 2015 Nov;139(11):1441-5. doi: 10.5858/arpa.2014-0454-OA. PMID 26516941
- [Background] Rozen P, Comaneshter D, Levi Z, Hazazi R, Vilkin A, Maoz E, Birkenfeld S, Niv Y. Cumulative evaluation of a quantitative immunochemical fecal occult blood test to determine its optimal clinical use. Cancer. 2010 May 1;116(9):2115-25. doi: 10.1002/cncr.25012. PMID 20186820
- [Derived] Daly JM, Xu Y, Crockett SD, Hoffman RM, Levy BT. Is Cognitive Impairment Associated with Inadequate Bowel Preparation for Colonoscopy? J Am Board Fam Med. 2025 Sep 15;38(3):423-430. doi: 10.3122/jabfm.2024.240338R1. PMID 40789626
- [Derived] Levy BT, Xu Y, Daly JM, Hoffman RM, Dawson JD, Shokar NK, Zuckerman MJ, Molokwu J, Reuland DS, Crockett SD. Comparative Performance of Common Fecal Immunochemical Tests : A Cross-Sectional Study. Ann Intern Med. 2024 Oct;177(10):1350-1360. doi: 10.7326/M24-0080. Epub 2024 Sep 3. PMID 39222513
- [Derived] Daly JM, Xu Y, Crockett SD, Schmidt ME, Kim P, Levy BT. Clock-Drawing Test as a Screening Tool for Cognitive Impairment Associated With Fecal Immunochemical Test Collection Errors. Ann Fam Med. 2022 Sep-Oct;20(5):452-459. doi: 10.1370/afm.2855. PMID 36228064
- [Derived] Levy BT, Daly JM, Xu Y, Crockett SD, Hoffman RM, Dawson JD, Parang K, Shokar NK, Reuland DS, Zuckerman MJ, Levin A. Comparative effectiveness of five fecal immunochemical tests using colonoscopy as the gold standard: study protocol. Contemp Clin Trials. 2021 Jul;106:106430. doi: 10.1016/j.cct.2021.106430. Epub 2021 May 8. PMID 33974994

DOCUMENTS (1):
  • Informed Consent Form (2021-05-07): https://cdn.clinicaltrials.gov/large-docs/98/NCT03264898/ICF_000.pdf